CLINICAL TRIAL: NCT02027688
Title: Feeding Progression in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Sara DeMauro, MD, MSCE, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 819247
Record Dates: First submitted 2013-12-31; First posted 2014-01-06 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Infant, Premature, Diseases; Feeding Behavior; Feeding Patterns
Keywords: Oral feeding; Premature; Infants; Neonatal Intensive Care Unit
MeSH Terms: conditions — Infant, Premature, Diseases; Feeding Behavior; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Every 6 hour Feeding Schedule (Active Comparator): Infants in this arm will be offered oral feedings every 6 hours if they are safe and ready to feed by mouth.
  Interventions: Other: q6 hour oral feeding schedule
- Every 3 Hour Oral Feeding (Active Comparator): Infants in this arm will be offered oral feedings every 3 hours if they are safe and ready to feed by mouth.
  Interventions: Other: q3 hour oral feeding schedule

INTERVENTIONS:
Other: q6 hour oral feeding schedule — The intervention is the schedule under which stable infants are offered oral feeding attempts: every 6 hours.
  Arms: Every 6 hour Feeding Schedule
Other: q3 hour oral feeding schedule — The intervention is the schedule under which stable infants are offered oral feeding attempts: every 3 hours.
  Arms: Every 3 Hour Oral Feeding

SUMMARY:
Preterm infants face many feeding challenges during hospitalization which can prolong hospitalization, raise parental anxiety and can lead to medical instability. The Feeding Progression study will randomize preterm infants to one of two currently accepted oral feeding schedules; oral feed attempts every 3 hours or every 6 hours. The study will collect data on oral feeding success, milk transfer, sucking strength, growth and medical complications.

DETAILED DESCRIPTION:
Preterm infants are at high risk for feeding issues. Feeding difficulties lead to prolonged hospitalization, increase medical complications and raise parental anxiety. The transition from tube feeding to oral feeding is an especially important step in a preterm infant's early life. Currently, there is limited evidence to guide this transition. There are two commonly used schedules for transitioning preterm infants to oral feeding: an every 6 hour schedule and an every 3 hour schedule. However, there is currently no evidence to guide providers in their choice of oral feeding schedule.

The primary objective of this study is to explore whether an every 6 (q6) hour oral feeding schedule will improve time to full oral feedings as compared to an every 3 (q3) hour oral feeding schedule. The secondary objectives are to test whether every 6 hour feeding allows for improved medical stability and oral-motor coordination as compared to the other commonly used q3 hour schedule. Each infant will be randomly assigned to a q6 hour or q3 hour oral feeding schedule. Data on oral feeding progression, respiratory status and oral motor proficiency will be collected and compared. The study will collect data on how long it takes each infant to get to full oral feeds, respiratory status throughout their time of oral feeding, whether there were any episodes of medical complications, measures of oral motor feeding skills, and the time to discharge from the hospital. This study is a crucial first step towards determining which feeding schedule is optimal for preterm infants to ensure timely attainment of full oral feeds and hospital discharge without compromising medical stability.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 23 0/7-33 0/7 weeks
* Eligible for oral (PO) feeding as determined by the attending Neonatologist

Exclusion Criteria:

* Infants with major congenital malformations
* Infants with chromosomal defects
* Diagnosis of Neonatal Abstinence Syndrome or opiate withdrawal
* Grade 3 or 4 Intraventricular Hemorrhage

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to full oral feeds | 38 weeks gestation on average
  Assess the relationship between feeding schedule and time to reach full oral feeds in preterm infants.

SECONDARY OUTCOMES:
Time to discharge | 40 weeks gestation on average
  Assess the relationship between feeding schedule and overall length of hospitalization.
Medical Complications | 38 weeks gestation on average
  Explore the relationship between feeding schedule and medical complications including apnea of prematurity, bronchopulmonary dysplasia, episodes of suspected sepsis, feeding intolerance and physiologic instability during the time of oral feeds.
Growth | 40 weeks gestation on average
  Assess the growth during the period of time from initiation of oral feeds to reaching complete oral feeds.
Feeding skills | 40 weeks gestation on average
  Assess feeding competence and sucking skills from initiation of feeds through discharge on full oral feeds.

CONTACTS AND LOCATIONS:
Overall Officials: Sara B DeMauro, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania